CLINICAL TRIAL: NCT03914742
Title: Phase I/II Study of BGB-290 With Temozolomide in Recurrent Gliomas With IDH1/2 Mutations
Brief Title: BGB-290 and Temozolomide in Treating Patients With Recurrent Gliomas With IDH1/2 Mutations
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH); BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABTC-1801; UM1CA137443 (NIH)
Record Dates: First submitted 2019-04-11; First posted 2019-04-16 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: IDH1 Mutation; IDH2 Mutation; Recurrent Glioblastoma; Recurrent WHO Grade II Glioma; Recurrent WHO Grade III Glioma
MeSH Terms: conditions — Glioblastoma | interventions — pamiparib; Temozolomide

STUDY DESIGN:
Intervention Model Description: Phase 1: BGB-290 in combination with TMZ in patients w/ IDH1/2-mutant WHO grade II-IV recurrent glioma: Phase 2: Grade II-III patients in will be stratified into 2 arms based on the timing of prior alkylator chemotherapy exposure; a third arm will include the subset of glioblastoma (grade IV) patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Phase 1: Dose Finding (Experimental): Recurrent IDH1/2-mutant grade II-III glioma: BGB290: Days 1-28, 60 mg PO BID TMZ: Days 1-28, 20 QD starting dose
  TMZ de-escalated treatment schedule if necessary (days 1-21; days 1-14; days 1-7) BGG held constant at 60mg PO BID
  Interventions: Drug: PARP Inhibitor BGB-290; Drug: Temozolomide
- Phase 2: Arm A Alkylator-resistant (Experimental): Grade II-III: Recurrent IDH1/2-mutant glioma (WHO grades II/III) who have failed TMZ AND another alkylator
  BGB290 + TMZ at dose combination established in Phase 1
  Interventions: Drug: PARP Inhibitor BGB-290; Drug: Temozolomide
- Phase 2: Arm B NOT Alkylator-resistant (Experimental): Grade II-III:Recurrent IDH1/2-mutant glioma (WHO grades II/III) Failed TMZ OR another alkylator;
  >/=12 months since last treatment
  BGB290 + TMZ at dose combination established in Phase 1
  Interventions: Drug: PARP Inhibitor BGB-290; Drug: Temozolomide
- GBM Arm (Experimental): Exploratory grade IV patients only BGB290 at Ph II dose for 7 days pre-surgery Progressed following RT + Chemo
  Interventions: Drug: PARP Inhibitor BGB-290; Drug: Temozolomide
- Surgical Arm (Experimental): Recurrent IDH1/2-mutant glioma (WHO grade II-IV) eligible for re-resection BGB-290: 60mg PO BID for 6 days AND day once day of surgery (day 7)
  Interventions: Drug: PARP Inhibitor BGB-290; Drug: Temozolomide; Procedure: Therapeutic Conventional Surgery

INTERVENTIONS:
Drug: PARP Inhibitor BGB-290 — Given PO
  Other Names: BGB-290, PARP, Inhibitor BGB-290
Drug: Temozolomide — Given PO
  Other Names: Temodar, Methazolastone
Procedure: Therapeutic Conventional Surgery — resection surgery
  Arms: Surgical Arm

SUMMARY:
This phase I/II trial studies the side effects and how well BGB-290 and temozolomide work in treating patients with gliomas (brain tumors) with IDH1/2 mutations that have come back. BGB-290 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving BGB-290 and temozolomide may work better in treating patients with recurrent gliomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

(Phase I) I. Determine the safety and tolerability of the combination of PARP inhibitor BGB-290 (BGB-290) and temozolomide (TMZ) in patients with recurrent IDH1/2 mutant glioma, including the maximum tolerated dose (MTD) and characterization of dose-limiting toxicities (DLTs) in the Phase I portion.

(Phase II) II. Determine the overall response rate of BGB-290 with TMZ in patients with recurrent IDH1/2-mutant gliomas that have progressed on TMZ and another alkylator (Arm A) in the Phase II portion.

III. Determine the overall response rate of BGB-290 with TMZ in patients with recurrent IDH1/2-mutant glioma that have failed one alkylator with >= 12 months since last treatment (Arm B) in the Phase II portion.

SECONDARY OBJECTIVES:

I. Determine the progression-free survival (PFS) and overall survival (OS) after treatment with BGB-290 and TMZ in recurrent IDH1/2-mutant gliomas in Arms A and B.

II. Determine the duration of response to therapy in recurrent IDH1/2-mutant glioma.

III. Confirm the safety and tolerability of BGB-290 in combination with TMZ.

EXPLORATORY OBJECTIVES:

I. Assess tumor response rates, PFS, and OS in patients with World Health Organization (WHO) grade IV glioblastoma (GBM) treated with BGB-290 and TMZ.

II. Assess the mutational landscape via whole-exome sequencing (WES). III. Assess gene expression patterns using ribonucleic acid (RNA) sequencing (RNAseq).

IV. Assess the methylation profiling with Infinium methylation assays. V. Quantify 2-hydroxyglutarate (2HG) in archival formalin-fixed paraffin-embedded (FFPE) specimens via liquid chromatography mass spectrometry (LC-MS) detection and correlate with treatment response.

VI. Correlate response with 2HG levels, somatic alterations, gene expression/methylation patterns in FFPE tumor tissue.

VII. Assess tumor tissue BGB-290 levels, 2HG, and PolyADP-ribosylation (PARylation) in a patient subset treated with drug prior to re-resection.

VIII. Evaluate changes in tumor growth rate in subjects with non-enhancing glioma based on fluid attenuated inverse recovery (FLAIR) tumor volume measurements of serial MRI exams.

IX. Assess if change in tumor growth rate (based on FLAIR tumor volume) in subjects with non-enhancing glioma before and after treatment is associated with progression by Response Assessment in Neuro-Oncology for Low Grade Gliomas (RANO LGG; phase II patients only) or survival.

OUTLINE: This is a phase I, dose de-escalation study of temozolomide followed by a phase II study.

PHASE I: Patients receive PARP inhibitor BGB-290 orally (PO) twice daily (BID) on days 1-28 and temozolomide PO once daily (QD) on days 1-28, 1-21, 1-14, or 1-7. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

SURGICAL PORTION: 10 patients eligible for re-resection at the time of recurrence receive PARP inhibitor BGB-290 PO BID on days 1-6 and QD on day 7 (the morning of surgery). Within 45 days after surgery, patients receive PARP inhibitor BGB-290 PO BID on days 1-28 and temozolomide on the schedule established in Phase I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PHASE II: Patients receive PARP inhibitor BGB-290 PO BID on days 1-28 and temozolomide PO QD on the schedule established in Phase I. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days, every 2 months for 2 years, then every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* PHASE I: Patients must have histologically confirmed WHO grade II-III glioma that is progressive or recurrent following at least one prior chemotherapy regimen plus or minus radiation therapy regimen or (b) Grade IV disease in their recurrent resection or biopsy specimen or (c) Grade IV glioma at initial diagnosis, with recurrent disease. Phase I patients may have failed an unlimited number of prior systemic regimens.
* PHASE II: Patients must have histologically confirmed WHO grade II-IV glioma that is progressive or recurrent following therapy:

  * Arm A patients must have WHO grade II-III glioma and have failed TMZ and another alkylator (e.g., carmustine, lomustine, procarbazine). Patients in Arm A may have failed an unlimited number of prior systemic regimens. Prior radiotherapy (RT) is not required for eligibility. There is no minimum time from the last antineoplastic treatment, except to allow for recovery: three weeks from last dose of TMZ and six weeks from last dose of nitrosourea.
  * Arm B patients must have WHO grade II-III glioma and have experienced tumor progression after TMZ or another alkylator (maximum one prior chemotherapy regimen), and have gone >= 12 months since last treatment (chemotherapy or RT). Prior radiation therapy (RT) is allowed but not mandated.
  * GBM Arm patients must have WHO grade IV glioblastoma following radiotherapy (45-60 gray [Gy] in 1.8-2.0 Gy fractions) plus chemotherapy and may have failed an unlimited number of prior systemic regimens.
  * Surgical portion patients must have histologically confirmed WHO grade II-IV glioma that is progressive or recurrent following therapy and must be undergoing repeat surgery that is clinically indicated as determined by their care providers. Surgical Portion patients may have had an unlimited number of prior therapy regimens.
  * Recurrence in non-enhancing tumors will be defined as 25% or more increase in bi-dimensional product of FLAIR signal abnormality (measurable disease) per the low-grade glioma (LGG) RANO criteria. Contrast-enhancing tumors with measurable enhancing targets will be defined as recurrent based on standard RANO criteria.
  * Patients with recurrent glioma < 12 weeks after completion of radiotherapy must have new enhancement outside of the RT field (beyond the high-dose region or 80% isodose line), or evidence of viable tumor on histopathologic sampling.
* PHASE I AND PHASE II: Patients must have available at least 3 prior full sets of magnetic resonance imaging (MRI) scans (not including screening), each separated by at least 2 months.
* Patients must have IDH1/2-mutant glioma. IDH1/2-mutation status can be confirmed by immunohistochemistry (IHC) or direct deoxyribonucleic acid (DNA) sequencing, provided that it is performed in a Clinical Laboratory Improvement Amendments/College of American Pathologists (CLIA/CAP)-certified laboratory. IDH1/2 mutations must be associated with neomorphic activity of the encoded proteins (i.e. IDH1 R132, IDH2 R172, IDH2 R140, IDH1 R100, IDH1 G97, IDH1 Y139).
* Patients must have archival formalin-fixed paraffin-embedded (FFPE) specimens and mutations will be verified centrally, although this will not preclude patients with appropriate documentation of IDH1/2-mutant status from trial enrollment. Patients must have a tumor tissue form indicating availability of archived tissue from a previous surgery, completed and signed by a pathologist; sites must agree to provide this form within 14 days after treatment start.
* Patients must have measurable (defined by at least 1 cm x 1 cm) contrast-enhancing disease or measurable abnormal T2/FLAIR hyperintensity indicative of tumor by MRI imaging within 21 days of starting treatment.
* Patients must have documented molecular 1p/19q and MGMT testing. If either of these studies has not been performed previously, they can be done prior to enrollment.
* Patients must be able to undergo MRI of the brain with gadolinium. Patients must be maintained on a stable or decreasing dose of corticosteroid regimen (no increase for 5 days) prior to this baseline MRI.
* Patients must have recovered from severe toxicity of prior therapy. The following intervals from previous treatments are required to be eligible:

  * 12 weeks from the completion of radiation
  * 6 weeks from a nitrosourea chemotherapy
  * 3 weeks from a non-nitrosourea chemotherapy
  * 4 weeks from any investigational (not Food and Drug Administration [FDA]-approved) agents
  * 2 weeks from administration of a non-cytotoxic, FDA-approved agent (e.g., erlotinib, hydroxychloroquine, etc.).
* Patients must have a Karnofsky performance (KPS) status >= 60% (i.e. the patient must be able to care for himself/herself with occasional help from others).
* Absolute neutrophil count >= 1,500/ uL.
* Platelets >= 100,000/ uL.
* Hemoglobin >= 9 g/dL.
* Total bilirubin =< institutional upper limit of normal.
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 4 × institutional upper limit of normal.
* Creatinine =< institutional upper limit of normal OR creatinine clearance >= 60 ml/min/1.73m^2 for patients with creatinine levels above institutional normal.
* Activated partial thromboplastin time (APTT) or PTT =< 1.5 × institutional upper limit of normal.
* Patients must be able to provide written informed consent.
* Women of childbearing potential must have a negative serum pregnancy test prior to study start. Women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and through 4 months after the last dose of study drug. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and through 4 months after completion of BGB-290 or temozolomide administration.
* Patients must have no concurrent malignancy except curatively treated basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix, breast, or bladder. Patients with prior malignancies must be disease-free for >= 5 years.
* Patients must be able to swallow tablets and capsules.

Exclusion Criteria:

* Patients receiving any other investigational agents are ineligible.
* Patients previously treated with a small molecule inhibitor of mutant IDH1/2 proteins are ineligible.
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to BGB-290 are ineligible.
* Patients who have received bevacizumab within the last 6 months are ineligible.
* Patients with a known hypersensitivity to TMZ are ineligible.
* Patients who have received a PARP inhibitor previously are excluded.
* Patients on enzyme-inducing anti-epileptic drugs (EIAED) are not eligible for treatment on this protocol. Patients may be on non-enzyme inducing anti-epileptic drugs or not be taking any anti-epileptic drugs. Patients previously treated with EIAEDs may be enrolled if they have been off the EIAED for 10 days or more prior to the first dose of BGB-290.
* Patients who have not recovered to < Common Terminology Criteria for Adverse Events (CTCAE) grade 2 toxicities apart from alopecia related to prior therapy are ineligible.
* Patients with uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, clinically significant cardiac disease, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements, are ineligible.
* Pregnant women are excluded from this study because the effects of BGB-290 on a fetus are unknown. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with BGB-290, breastfeeding should be discontinued if the mother is treated with BGB-290.
* Human immunodeficiency virus (HIV)-positive patients on combination antiretroviral therapy are ineligible due to potential drug-drug interactions with BGB-290.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2020-02-16 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ranjit Bindra, MD, Study Chair — ABTC/Yale University; David Schiff, MD, Study Chair — ABTC/University of Virginia
Locations (12):
- United States (12):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - University of California, Los Angeles, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Josephine Ford Cancer Center at Henry Ford Hospital, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Hillman Cancer Center at University of Pittsburgh Cancer Institute, Pittsburgh, Pennsylvania
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment started Feb 2020 & the last patient enrolled 4/4/22. The trial terminated early due to mandated closed to accrual and treatment on October 31 2023. The final clinical data includes a total of 67 subjects enrolled and 66 evaluable. Due to mandated closure of treatment and follow-up on 10/31/23, many patients were moved to compassionate use and dealth dates post 10/31/23 could not be collected or confirmed. The termination of the trial is considered an administrative termination.
Pre-assignment Details: 67 patients signed consent, however, 1 patient in the Phase 1 Dose Finding, never started treatment before they withdrew, hence 66 evaluable patients.
Groups:
- Phase 1: Dose Finding: Recurrent IDH1/2-mutant grade II-III glioma: BGB290: Days 1-28, 60 mg PO BID TMZ: Days 1-28, 20 QD starting dose
  PARP Inhibitor BGB-290 60mg BID: Given PO
  Temozolomide 20mg QD: Given PO
- Phase 2: Arm A Alkylator-resistant: Grade II-III: Recurrent IDH1/2-mutant glioma (WHO grades II/III) who have failed TMZ AND another alkylator
  PARP Inhibitor BGB-290 60mg BID: Given PO
  Temozolomide 20mg QD: Given PO
- Phase 2: Arm B NOT Alkylator-resistant: Grade II-III:Recurrent IDH1/2-mutant glioma (WHO grades II/III) Failed TMZ OR another alkylator;
  >/=12 months since last treatment
  PARP Inhibitor BGB-290 60mg BID: Given PO
  Temozolomide 20mg QD: Given PO
- GBM Arm: Exploratory grade IV patients only Progressed following RT + Chemo
  PARP Inhibitor BGB-290 60mg BID: Given PO
  Temozolomide 20mg QD: Given PO
- Surgical Arm: Recurrent IDH1/2-mutant glioma (WHO grade II-IV) eligible for re-resection BGB-290: 60mg PO BID for 6 days AND day once day of surgery (day 7)
  post surgery PARP Inhibitor BGB-290 60mg BID: Given PO
  Temozolomide 20mg QD: Given PO
  Therapeutic Conventional Surgery: resection surgery
Period: Overall Study
Arm/Group | Phase 1: Dose Finding | Phase 2: Arm A Alkylator-resistant | Phase 2: Arm B NOT Alkylator-resistant | GBM Arm | Surgical Arm
Started | 7 | 15 | 24 | 10 | 10
Completed | 7 | 15 | 24 | 10 | 10
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: In the Phase 1: Dose Finding arm, 8 patients signed consent, however 1 patient withdrew prior to starting treatment. Hence a total of 7 patients evaluable for the Phase 1 portion of the study
Groups:
- GBM Arm: Exploratory grade IV patients only progressed following RT and TMZ
  PARP Inhibitor BGB-290 60mg BID: Given PO
  Temozolomide 20mg QD: Given PO
- Total: Total of all reporting groups
Arm/Group | Phase 1: Dose Finding | Phase 2: Arm A Alkylator-resistant | Phase 2: Arm B NOT Alkylator-resistant | GBM Arm | Surgical Arm | Total
Number analyzed (Participants) | 7 | 15 | 24 | 10 | 10 | 66
Age, Continuous [Median (Full Range); unit: years] | 45.2 [25.4 to 54.6] | 42.7 [35.9 to 58.4] | 45.5 [22.2 to 68.6] | 35.9 [23.5 to 72.9] | 46.7 [32.8 to 66.9] | 44.5 [22.2 to 72.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 12 | 5 | 4 | 29
  Male | 4 | 10 | 12 | 5 | 6 | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 2 | 1 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 0 | 1 | 2
  White | 6 | 12 | 21 | 7 | 8 | 54
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 1 | 2 | 1 | 6
Number of Relapes [Median (Full Range); unit: relapses] | 3 [1 to 4] | 2 [2 to 3] | 1 [1 to 3] | 2 [1 to 7] | 2 [1 to 2] | 1 [1 to 7]
Molecular Markers (1p/19q) [Count of Participants; unit: Participants] — molecular markers determined by testing tumor tissue
  Participants
    Co-deleted | 2 | 9 | 18 | 1 | 3 | 33
    intact | 4 | 5 | 5 | 8 | 7 | 29
    19q-deleted only | 1 | 0 | 1 | 1 | 0 | 3
    Not Done | 0 | 1 | 0 | 0 | 0 | 1
MGMT gene (Methylated) [Count of Participants; unit: Participants] — MGMT (O-6-methylguanine methyl transferase) is a gene.
  Participants | 1 | 9 | 19 | 6 | 5 | 40
Type of Surgical Proceedure [Count of Participants; unit: Participants]
  Gross Total Resection | 4 | 9 | 9 | 7 | 5 | 34
  Subtotal Resection | 2 | 6 | 14 | 2 | 4 | 28
  Biopsy | 1 | 0 | 1 | 1 | 1 | 4
Karnosky Performance Status (KPS) [Median (Full Range); unit: units on a scale] — Higher score better 100 normal no complaints/disease 90 capable normal activity few symptoms/disease 80 normal activity, some difficulty some symptoms/signs 70 caring for self not capable normal activity/work 60 requiring some help can take care of most personal requirements 50 requires help often requires frequent medical care 40 disabled requires special care/help 30 severely disabled hospital admission indicated but no risk of death 20 very ill urgently requiring admission requires supportive measures/treatment 10 moribund rapidly progressive fatal disease processes 0 death
  units on a scale | 90 [70 to 100] | 80 [70 to 100] | 90 [60 to 100] | 90 [70 to 100] | 90 [60 to 100] | 90 [60 to 100]

OUTCOME MEASURES:

1. Primary Outcome: Participants With Dose Limiting Toxicity (DLT) Rate Less Than or Equal to 33% (Dose Level 1)
Description: DLTS defined as the combination regimen that yields a dose limiting toxicity (DLT) rate less than, or equal to 33%. A DLT is defined as a clinically significant adverse event or abnormal laboratory value assessed as unrelated to disease progression, intercurrent illness, or concomitant medications and meets any of the criteria below. Any DLT must be a toxicity considered at least possibly related to pamiparib (BGB-290) or TMZ.
Time Frame: up to 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Dose Level 1 (Starting Dose): Recurrent IDH1/2-mutant grade II-III glioma: BGB290: Days 1-28, 60 mg PO BID TMZ: Days 1-28, 20mg QD
  PARP Inhibitor BGB-290: Given PO
  Temozolomide: Given PO
Arm/Group | Dose Level 1 (Starting Dose)
Number analyzed (Participants) | 7
Participants
  DLT rate >33% | 0
  DLT rate <33% | 7

2. Primary Outcome: Maximum Tolerated Dose
Description: Patients treated with TMZ 20mg Days 1-28, highest dose level/schedule. If DTL observed, dose level/schedule will de-escalated treatment schedule if necessary (days 1-21; days 1-14; days 1-7) BGG held constant at 60mg PO BID
Time Frame: up to 28 days
Measure: Count of Participants; unit: Participants
Groups:
- Phase 1: Dose Finding: Recurrent IDH1/2-mutant grade II-III glioma: BGB290: Days 1-28, 60 mg PO BID TMZ: Days 1-28, 20 QD starting dose
  TMZ de-escalated treatment schedule if necessary (days 1-21; days 1-14; days 1-7) BGG held constant at 60mg PO BID
  PARP Inhibitor BGB-290: Given PO
  Temozolomide: Given PO
Arm/Group | Phase 1: Dose Finding
Number analyzed (Participants) | 7
Participants
  TMZ 20mg 1-28 Days | 7
  TMZ 20mg 1-21 Days | 0
  TMZ 20mg 1-14 Days | 0

3. Primary Outcome: Phase II: Overall Best Response Rate for Arm A and Arm B
Description: Number of participants with response as defined by Response Assessment in Neuro-oncology (RANO) criteria: Complete Response (CR)= no change in size of T1-gadolinium-enhancing (T1-Gd+) disease, stable or reduced T2/FLAIR signal, no new lesion, no corticosteroid use, and stable or improved clinical status; Partial Response (PR)= ≥50% change in size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Stable Disease (SD)= <50% reduction to <25% increase size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Progressive Disease (PD)= ≥25% increase size of T1-Gd+ disease, or increased T2/FLAIR signal, or presence of new lesion, or worsening clinical status.
Time Frame: up to 2 years
Measure: Number; unit: participants
Arm/Group | Phase 2: Arm A Alkylator-resistant | Phase 2: Arm B NOT Alkylator-resistant
Number analyzed (Participants) | 15 | 24
participants
  Complete Response | 0 | 0
  Partial Response | 0 | 1
  Stable disease | 9 | 18
  Progressive Disease | 5 | 1
  Not Adequately Assessed | 1 | 4

4. Secondary Outcome: Phase II: Progression-free Survival (PFS) in Arm A and Arm B
Description: Time from date of treatment start to date of initial scan indicating progression
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Arm A Alkylator-resistant | Phase 2: Arm B NOT Alkylator-resistant
Number analyzed (Participants) | 15 | 24
months | 5.9 [1.2 to 14.8] | 9.7 [5.7 to 21.7]

5. Secondary Outcome: Phase II: Overall Survival (OS) for Arm A and Arm B
Description: Median time from start date of treatment to date of death
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Phase 2: Arm A Alkylator-resistant | Phase 2: Arm B NOT Alkylator-resistant
Number analyzed (Participants) | 15 | 24
months | 26.1 [6.0 to NA] — Results for the outer bounds were not reached for this outcome measure. Overall Survival data were not all mature for reporting, the trial was closed early due to the mandated closure of the ABTC consortium by NCI/CTEP to explore new designs for CNS Consortiums | NA [22 to NA] — Results for the outer bounds were not reached for this outcome measure. Overall Survival data were not all mature for reporting, the trial was closed early due to the mandated closure of the ABTC consortium by NCI/CTEP to explore new designs for CNS Consortiums

6. Secondary Outcome: Duration of Response Phase 2
Description: Time from date of initial scan indicating complete or partial response to a date of the initial scan deemed tumor progression. Response is defined by RANO criteria as follows: Complete Response (CR)= no change in size of T1-gadolinium-enhancing (T1-Gd+) disease, stable or reduced T2/FLAIR signal, no new lesion, no corticosteroid use, and stable or improved clinical status; Partial Response (PR)= ≥50% change in size of T1-Gd+ disease, stable or reduced T2/FLAIR signal, no new lesion, stable or reduced corticosteroid use, and stable or improved clinical status; Progressive Disease (PD)= ≥25% increase size of T1-Gd+ disease, or increased T2/FLAIR signal, or presence of new lesion, or worsening clinical status.
Time Frame: up to 2 years
Measure: Number; unit: weeks
Arm/Group | Phase 2: Arm A Alkylator-resistant | Phase 2: Arm B NOT Alkylator-resistant
Number analyzed (Participants) | 15 | 24
weeks
  Duration of complete response (CR) | 0 | 0
  Duration of partial response (PR) | 0 | 10.9

ADVERSE EVENTS:
Time Frame: Start of treatment to 30 days post last dose. Approximately 2 years
Groups:
- Phase 1: Dose Finding: Recurrent IDH1/2-mutant grade II-III glioma: BGB290: Days 1-28, 60 mg PO BID TMZ: Days 1-28, 20 QD starting dose & MTD
  PARP Inhibitor BGB-290 60mg BID: Given PO
  Temozolomide 20mg QD: Given PO
Arm/Group | Phase 1: Dose Finding | Phase 2: Arm A Alkylator-resistant | Phase 2: Arm B NOT Alkylator-resistant | GBM Arm | Surgical Arm
All-Cause Mortality (participants affected / at risk) | 4/7 | 4/15 | 6/24 | 6/10 | 3/10
Serious Adverse Events (participants affected / at risk) | 1/7 | 0/15 | 2/24 | 1/10 | 3/10
Other Adverse Events (participants affected / at risk) | 7/7 | 15/15 | 24/24 | 10/10 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Finding (N=7) | Phase 2: Arm A Alkylator-resistant (N=15) | Phase 2: Arm B NOT Alkylator-resistant (N=24) | GBM Arm (N=10) | Surgical Arm (N=10)
Acute Kidney Injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 3 hospitalization
Alanine aminotransferase increase (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — ALT Grade 3 Hospitalized
Anemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 3 Hospitalization
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Grade 3 Hospitilaztion
headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Grade 3 Hospitalization
intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 3 Hospitalization
Lymphocyte count decrease (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Grade 3 and grade 4 Hospitalization
Neutrophile count decrease (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Grade 3 and 4 Hospitalization
Platelet count decrease (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Grade 3 and 4 Hospitalization
Renal calculi (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) — Grade 3 Hospitalization
White Blood Cell Count Decrease (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) — Grade 4 hospitalization
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase 1: Dose Finding (N=7) | Phase 2: Arm A Alkylator-resistant (N=15) | Phase 2: Arm B NOT Alkylator-resistant (N=24) | GBM Arm (N=10) | Surgical Arm (N=10)
Alanine aminotransferase increase (Investigations) | 1 (2) | 3 (6) | 6 (9) | 3 (3) | 1 (2)
Gastroesophageal Acid Reflux (Gastrointestinal disorders) | 3 (3) | 0 (0) | 0 (0) | 1 (2) | 0 (0) — Acid Reflux
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 6 (7) | 0 (0) | 0 (0) — loss of appetite
anemia (Blood and lymphatic system disorders) | 3 (11) | 11 (36) | 20 (219) | 8 (29) | 7 (27)
Aspartate aminotransferase increased (Investigations) | 1 (2) | 2 (2) | 3 (6) | 3 (10) | 0 (0)
Blood Bilirubin increase (Investigations) | 0 (0) | 0 (0) | 3 (8) | 0 (0) | 0 (0)
chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (3) | 1 (1) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 0 (0)
dizziness (Nervous system disorders) | 0 (0) | 2 (2) | 4 (4) | 2 (2) | 0 (0)
Fatigue (General disorders) | 4 (4) | 10 (16) | 14 (18) | 3 (3) | 3 (4)
flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 1 (2) | 2 (2) | 1 (1) | 0 (0) — General stomach issues
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (2)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphatemia (Metabolism and nutrition disorders) | 1 (5) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hypertension (Cardiac disorders) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Hypophosphatemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 3 (6) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lymphocyte count decreased (Investigations) | 4 (6) | 4 (15) | 13 (49) | 4 (18) | 4 (9)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 3 (3) | 2 (3) | 16 (21) | 3 (3) | 4 (5)
Neutrophil count decreased (Investigations) | 4 (24) | 8 (42) | 17 (152) | 6 (21) | 5 (25)
Platelet count decreased (Investigations) | 2 (8) | 8 (22) | 16 (60) | 8 (34) | 6 (19)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
vomiting (Gastrointestinal disorders) | 1 (2) | 2 (2) | 3 (5) | 0 (0) | 2 (2)
Weight loss (Investigations) | 2 (2) | 0 (0) | 2 (2) | 1 (2) | 0 (0)
White blood cell decreased (Investigations) | 4 (28) | 9 (63) | 18 (236) | 7 (38) | 6 (28)

LIMITATIONS AND CAVEATS:
This study did finish enrollment for all arms (67 patients) however, due to mandated shut down by NCI/CTEP of our ABTC Consortium not all patients were able to complete treatment on study and/or have PFS or OS mature to use for outcomes (statistics). Additionally, many of the exploratory endpoints were not completed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-07-07): https://cdn.clinicaltrials.gov/large-docs/42/NCT03914742/Prot_SAP_000.pdf